CLINICAL TRIAL: NCT04521959
Title: The Effect Of Blood Flow Restrıcted Resistive And Aerobic Exercises in Chronic Obstructive Pulmonary Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ahmet Gunes, PhD Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: istanbul medipol university
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Copd
Keywords: COPD, blood flow restriction, exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Two randomized controlled intervention groups will be formed.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 40 COPD patients will be randomised divided into two equal groups according to age, gender and disease severity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restricted Aerobic and Resistance Exercise Group (Active Comparator): kan akımı kısıtlanarak.direnç ve bisikletle aerobik egzersiz uygulanacak
  Interventions: Procedure: Blood flow restricted and normal aerobic exercise and resistance exercise
- Normal aerobik ve direnç egzersiz grubu (Active Comparator): Normal şartlarda aerobik ve direnç egzersizi uygulanacak
  Interventions: Procedure: Blood flow restricted and normal aerobic exercise and resistance exercise

INTERVENTIONS:
Procedure: Blood flow restricted and normal aerobic exercise and resistance exercise — Interventions of the same duration and intensity will be applied to two groups.

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) classified by a pulmonologist in accordance with the GOLD criteria will be randomly divided into 2 groups.

The first group (n = 20) was accompanied by blood flow restriction (CAC), 3 times a week, 8 weeks, 1RMx 30% intensity, 10 repetitions, 3 sets, 30 seconds rest interval, progressive resistance exercise (PRE) and after 5 minutes of rest by cycling. Progressive aerobic exercise (AE) (BFR PRE + AE group) in the target heart rate range of 50-80% intensity will be applied to the second group (n = 20), PRE and AE (PRE + AE group) performed at the same intensity and duration without BFR.

DETAILED DESCRIPTION:
Determination of application groups: Patients with chronic obstructive pulmonary disease (COPD) classified by a pulmonologist in accordance with the GOLD criteria will be randomly divided into 2 groups and application groups will be determined.

Applications to be made:

The first group (n = 20) accompanied by BFR; Progressive resistance training (RT) 3 times a week, 1RMx 30% intensity, 10 repetitions, 3 sets, 30 seconds rest interval, and cycling after 5 minutes rest, progressive aerobic training (AT)in the target heart rate range of 40-80% intensity will be applied.

To the second group (n = 20) without BFR; 3 times a week, 8 weeks, 1RMx 30% intensity, 10 repetitions, 3 sets, 30 seconds of rest interval, and after 5 minutes of rest will be applied in the target heart rate range of 40-80%, which is done by cycling.

Calculation of 1RM: Epley formula will be used in the calculation. According to this; 1 RM = (1 + .0333 x number of repetitions) x weight removed.

Progress in resistance exercise; According to the modified borg scale (MBS), the amount of the lifted weight calculated on the basis of the increase in the 1RM value measured in every three consecutive sessions will be provided by increasing the amount of weight, on the condition that it remains between 4-6 intensity.

This too; It will be calculated from the formula "Target heart rate = (Maximal heart rate-resting heart rate) x% desired intensity ratio + resting heart rate".

The target occlusion amount in the lower extremity will be calculated by calculating 45% of the complete occlusion rates reported by Michael et al. The proximal border of the thigh cuffs in the BFR group will be tied at the level of the gluteal lines on both sides.

Exercise tolerance and dyspnea condition; Measurement properties in COPD will be evaluated using a modified Borg scale (MBS), which has well-defined characteristics. Individuals will use bronchodilators approved by their physician before each trial and continue drug therapy throughout the study.

The target aerobic exercise intensity will be reached in the last minute of the first five-minute warm-up period by maintaining a 4-6 feeling of dyspnea in the MBS, by increasing pedal resistance and speed. The intensity increase will be increased by 5% for each subsequent session and the target heart rate will be limited to 80%. In case of extreme shortness of breath, the intensity of exercise will be reduced down to the resting heart rate.

In case of oxygen desaturation (85%) during interventions, the intervention will be suspended until the next session.

Aerobic exercise study protocol: warm-up at 50 RPM speed and lowest pedal resistance for the first 4 minutes, reaching the target exercise intensity range in the next 1 min, aerobic training at the target heart rate range and appropriate MBS for the next 20 minutes, the last 5 minutes It will be applied in the form of cooling. The duration will be reduced in case of extreme shortness of breath, fatigue and muscle pain due to increased exercise volume. The distance, calories, and maximum speed values measured during the first, 9 and 24 sessions will be recorded.

Before the study and at the end of the 8th week, oxidative stress markers (plasma protein carbonyl concentration, lipid hydroperoxides, total antioxidant capacity (TAK)), muscle damage status (creatine phosphokinase, myoglobin), anti-inflammatory response (interleukin 6 (IL-6), risk of venous thromboembolism and thrombus formation (D-dimer, thrombin-antithrombin 3 component (TAT), c-reactive protein (CRP), fibrinogen), body mass index, respiratory function tests (FEV1, FVC), oxygen saturation and heart rate ( pulse oximetry), six-minute walking test, and quality of life (SF-36) will be evaluated at least 6 hours prior to taking medication.

The change in the quadriceps muscle mass will be examined by a radiologist who is not involved in the study, by measuring the transverse and anteroposterior lengths of the relevant muscle using Toshiba aplio 300 brand ultrasound device.

Statistical evaluation of results: Paired t-test, repeated measurement analysis of variables (RMANOVA), Kolmogorov-Smirnov test, post hoc contrast analysis, bonferroni correction will be used in the statistical analysis of intervention results.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mild to severe COPD according to GOLD criteria in the age range of 40-78
* No drug change for at least 30 days
* Not participating in a structured activity program for at least six months
* Have the ability to cooperate.

Exclusion Criteria:

* Presence of any pathology that limits physical activity performance
* Presence of severe or unstable heart disease
* Presence of peripheral artery disease
* Being in an exacerbation period of the disease
* Presence of another active disease (rheumatic, oncological, traumatic etc.)
* Any neurological or orthopedic disease that prevents exercise

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since COPD affects male gender more, the number of male patients participating in the intervention is higher than female patients.
Enrollment: 40 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
FEV1/FVC rate | eight weeks
  respiratory function test
creatine kinase | eight weeks
  muscle breakdown marker
c reactive protein | eight weeks
  thrombus formation risk marker
d-dimer | eight weeks
  venous thromboembolism marker
total antioxidant status | eight weeks
  oxidative stress marker
total oxidant status | eight weeks
  oxidative stress marker
interleukin 6 | eight weeks
  inflammation marker
oxygen saturation | three times a week
  blood gas test
heart rate | three times a week
  for exercise dose determination
six minute walk test | eight weeks
  strength evaluation
ST george's respiratory questionnaire | eight weeks
  used to evaluate the effects of respiratory disease's symptoms and illness
quadriceps muscle diameter | eight weeks
  Measurement of change in muscle volume

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük Üniversitesi Araştırma Hastanesi Göğüs Hastalıkları Kliniği, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Nolan CM, Rochester CL. Exercise Training Modalities for People with Chronic Obstructive Pulmonary Disease. COPD. 2019 Dec;16(5-6):378-389. doi: 10.1080/15412555.2019.1637834. Epub 2019 Nov 4. PMID 31684769
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Background] Kacin A, Strazar K. Frequent low-load ischemic resistance exercise to failure enhances muscle oxygen delivery and endurance capacity. Scand J Med Sci Sports. 2011 Dec;21(6):e231-41. doi: 10.1111/j.1600-0838.2010.01260.x. Epub 2011 Mar 8. PMID 21385216
- [Background] Loenneke JP, Allen KM, Mouser JG, Thiebaud RS, Kim D, Abe T, Bemben MG. Blood flow restriction in the upper and lower limbs is predicted by limb circumference and systolic blood pressure. Eur J Appl Physiol. 2015 Feb;115(2):397-405. doi: 10.1007/s00421-014-3030-7. Epub 2014 Oct 22. PMID 25338316
- [Background] Wilson JM, Lowery RP, Joy JM, Loenneke JP, Naimo MA. Practical blood flow restriction training increases acute determinants of hypertrophy without increasing indices of muscle damage. J Strength Cond Res. 2013 Nov;27(11):3068-75. doi: 10.1519/JSC.0b013e31828a1ffa. PMID 23446173
- [Background] Berzosa C, Cebrian I, Fuentes-Broto L, Gomez-Trullen E, Piedrafita E, Martinez-Ballarin E, Lopez-Pingarron L, Reiter RJ, Garcia JJ. Acute exercise increases plasma total antioxidant status and antioxidant enzyme activities in untrained men. J Biomed Biotechnol. 2011;2011:540458. doi: 10.1155/2011/540458. Epub 2011 Mar 9. PMID 21436993
- [Background] Wilk M, Krzysztofik M, Gepfert M, Poprzecki S, Golas A, Maszczyk A. Technical and Training Related Aspects of Resistance Training Using Blood Flow Restriction in Competitive Sport - A Review. J Hum Kinet. 2018 Dec 31;65:249-260. doi: 10.2478/hukin-2018-0101. eCollection 2018 Dec. PMID 30687436